CLINICAL TRIAL: NCT06565312
Title: A Single Group Study to Evaluate the Effects of a Probiotic Vaginal Suppository on Vaginal Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20434
Record Dates: First submitted 2024-07-11; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Vaginal Health; Vaginal pH
Keywords: Vaginal suppository; Women's Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flora Power Probiotic Vaginal Suppository (Experimental): Participants will use the Flora Power suppository once daily at bedtime for 5 consecutive days when they feel they are experiencing any of the common signs of vaginal imbalance like vaginal malodor, vaginal irritation, and/or vaginal itching.
  Interventions: Dietary Supplement: Flora Power Probiotic Vaginal Suppository

INTERVENTIONS:
Dietary Supplement: Flora Power Probiotic Vaginal Suppository — The suppository contains Microcrystalline Cellulose, Ascorbic Acid, Vitamin C, Gelatin Capsule, Vaginal Probiotic Blend (Lactobacillus fermentum LF61, Lactobacillus acidophilus LA85, Lactobacillus plantarum Lp90), Magnesium Stearate, and Silicon Dioxide.

SUMMARY:
This is a virtual single-group clinical trial lasting 8 weeks to evaluate the effects of a probiotic vaginal suppository on vaginal health. Participants will use the Flora Power suppository daily for 5 consecutive days when experiencing common signs of vaginal imbalance. They will complete questionnaires and vaginal pH tests before and after product use.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth, aged 18+.
* Interested in maintaining a healthy vaginal environment.
* Experience common signs of vaginal imbalance (e.g., malodor, irritation).
* Willing to avoid other vaginal products and follow study protocol.

Exclusion Criteria:

* Recent surgeries or invasive treatments.
* Use of vaginal health products in the last 12 weeks.
* Allergies to product ingredients.
* Chronic health conditions impacting participation.
* Pregnant, breastfeeding, or trying to conceive.
* History of substance abuse or smoking.
* Currently participating in another clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Effect on Vaginal pH and Health | Baseline, Day 6 (24 hours after the last suppository insertion)
  Measure the change in vaginal pH levels with a test strip from baseline to 24 hours after the 5-day intervention period.
Effect on Vaginal pH and Health | Baseline, Day 6 (24 hours after the last suppository insertion)
  Measure the change in overall vaginal health from baseline to 24 hours after the 5-day intervention period with a questionnaire.

SECONDARY OUTCOMES:
Participant Perception of Vaginal Freshness and Odor | Baseline, Day 2, Day 5
  Evaluate participants' perceptions of the vaginal suppository's impact on vaginal freshness and odor, as well as the support of a calm, soothed, and balanced vaginal environment. This outcome measure is assessed with questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No